CLINICAL TRIAL: NCT06115824
Title: A Retrospective Case-control Study of Newly-diagnosed Primary Central Nervous System Lymphoma (PCNSL) Treated With Methotrexate (MTX)-Based Chemotherapy in Combination With Orelabrutinib
Brief Title: New-diagnosed PCNSL Treated With Methotrexate (MTX) and Orelabrutinib-based Regimen
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Tong Chen, MD, Prof., Huashan Hospital
Other Study IDs: KY2023-677
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Cohort A was the cohort of patients who received methotrexate-based chemotherapy alone
- Cohort B: cohort B was the cohort of patients who received methotrexate-based chemotherapy + orelabrutinib.
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — Combination of orelabrutinib on a methotrexate-based chemotherapy regimen with a starting dose of 150 mg/d
  Groups: Cohort B

SUMMARY:
This study was a single-centre, retrospective study that retrospectively collected first-line PCNSL patients receiving methotrexate-based chemotherapy ± orelabrutinib at Huashan Hospital of Fudan University. The study was divided into two retrospective cohorts, Cohort A was a cohort of patients receiving methotrexate-based chemotherapy alone, and Cohort B was a cohort of patients receiving methotrexate-based chemotherapy + orelabrutinib.

DETAILED DESCRIPTION:
The study was divided into two retrospective cohorts of approximately 35-40 patients each. Cohort A was the cohort of patients who received methotrexate-based chemotherapy alone, and cohort B was the cohort of patients who received methotrexate-based chemotherapy + orelabrutinib. Statistical analyses such as propensity score analysis (PSM) and inverse probability weighted (IPTW) analysis were performed, focusing on comparing and analysing the short-term efficacy data (ORR, CR) and long-term efficacy data (PFS, OS) of the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed primary central nervous system lymphoma
* Methotrexate-based chemotherapy ± orelabrutinib regimen as first-line treatment for patients

Exclusion Criteria:

* Patients receiving ≤2 cycles of treatment without efficacy evaluation
* Those with uncontrolled or significant cardiovascular disease, including: uncontrolled diabetes mellitus, severe cardiac, pulmonary, hepatic, renal insufficiency) and haematological, endocrine system lesions, history of other uncontrollable malignancies

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PCNSL is a rare and highly aggressive subtype of primary extranodal non-Hodgkin's lymphoma with a distinctive clinical presentation, and more than 95% of the pathological types are diffuse large B-cell lymphomas.The current National Comprehensive Cancer Network (NCCN) guidelines recommend first-line induction therapy with high-dose methotrexate (HD-MTX) in combination with rituximab, but long-term efficacy is still unsatisfactory, with 50% of patients relapsing at around 2 years
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of induction therapy, Cycle 6-8 (each cycle is 28 days)
  ORR is defined as the proportion of patients with a best response of CR, CRu or PR during induction therapy

SECONDARY OUTCOMES:
PFS | Up to 2 years
  Progression-free survival is calculated from the date of start of therapy until the date of first documented progress or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tong Chen, Principal Investigator — Huashan Hospital; Tong Chen, Study Director — Huashan Hospital
Locations (1):
- Department of Hematology, Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No